CLINICAL TRIAL: NCT05054127
Title: Clinical Characteristics And Outcome Of COVID-19 Infection In Patients With Chronic Respiratory Diseases.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madonna Youssef Roshdy Kelada, Madonna youssef roshdy kelada, Assiut University
Other Study IDs: COVID-19 and CRD
Record Dates: First submitted 2021-09-21; First posted 2021-09-23 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Chronic Respiratory Disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: foiiow up patients — observational study

SUMMARY:
1. To identify the pattern of presentation of COVID-19 in patients with chronic respiratory diseases
2. To asses the severity of COVID-19 in patients with chronic respiratory diseases
3. To identify the outcome of COVID-19 in patients with chronic respiratory diseases

DETAILED DESCRIPTION:
Genomes analysis reveal that SARS-CoV-2 presents unique features: optimal affinity for angiotensin converting enzyme 2 (ACE2) receptor and a polybasic cleavage site at the S1/S2 spike junction that determines infectivity and host range [3-4) Patients with SARS-CoV-2 infection may present symptoms ranging from mild to severe with a large portion of the population being asymptomatic carriers. The most common reported symptoms include fever (83%), cough (82%) and shortness of breath (31%) [5-6]. Patients suffering from chronic respiratory diseases (CRD) such as chronic respiratory failure, asthma, chronic obstructive pulmonary disease (COPD), interstitial lung diseases (ILD), pulmonary hypertension (PH), sarcoidosis or cystic fibrosis (CF), were immediately considered to be at risk of severe forms of COVID-19 [7]. Indeed, COVID-19 is responsible for various respiratory symptoms, from cough with dyspnea to acute respiratory distress syndrome (ARDS) in its most severe presentation [8-9]. In parallel, it has been shown that COVID-19 patients have an increased risk of venous thromboembolic disease [10]. There is concern that the respiratory complications of COVID-19 could be deleterious in patients with prior CRD. [11-12-13] During COVID-19 pandemic, studies mostly demonstrated that COPD was related with worse outcomes. There may be a few reasons why the course of COVID-19 in COPD patients has been worse. Firstly, COPD patients tend to be older and have more comorbidities which may increase COVID-19 severity [14]. Respiratory failure and hypoxemia, which are the most important causes of death in COVID-19 patients, are more common in COPD patients [15]. Although the exact mechanism of acute exacerbation of ILD is not fully understood, the current belief is that it can be caused by numerous triggers, including infection, or it can be idiopathic.(16) It is likely that respiratory infection with COVID-19 could trigger an exacerbation of underlying ILD and result in poor outcomes. There is similar concern regarding the possibility of exacerbation in patients with sarcoidosis, especially those with fibrotic manifestations.(17)

1. To identify the pattern of presentation of COVID-19 in patients with chronic respiratory diseases
2. To asses the severity of COVID-19 in patients with chronic respiratory diseases
3. To identify the outcome of COVID-19 in patients with chronic respiratory diseases

ELIGIBILITY:
Inclusion Criteria:

1. patients with chronic respiratory diseases diagnosed with covid-19 infection by PCR
2. Patients aged 18 years and above

Exclusion Criteria:

1. Patient aged below 18 years old.
2. Patients refuse to share in our study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with chronic respiratory diseases present with covid 19 infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
relation between covid 19 and patients with chronic respiratory diseases | Baseline
  pattern of presentation of COVID-19 in patients with chronic respiratory diseases 2-To asses the severity of COVID-19 in patients with chronic respiratory diseases 3-To identify the outcome of COVID-19 in patients with chronic respiratory diseases The pattern of presentation of COVID-19 in patients with chronic respiratory diseases The severity of COVID-19 in patients with chronic respiratory diseases The outcome of COVID-19 in patients with chronic respiratory diseases

REFERENCES:
- [Background] Cakir Edis E. Chronic Pulmonary Diseases and COVID-19. Turk Thorac J. 2020 Sep;21(5):345-349. doi: 10.5152/TurkThoracJ.2020.20091. Epub 2020 Sep 1. PMID 33031727
- [Background] Alqahtani JS, Oyelade T, Aldhahir AM, Alghamdi SM, Almehmadi M, Alqahtani AS, Quaderi S, Mandal S, Hurst JR. Prevalence, Severity and Mortality associated with COPD and Smoking in patients with COVID-19: A Rapid Systematic Review and Meta-Analysis. PLoS One. 2020 May 11;15(5):e0233147. doi: 10.1371/journal.pone.0233147. eCollection 2020. PMID 32392262
- [Background] Poissy J, Goutay J, Caplan M, Parmentier E, Duburcq T, Lassalle F, Jeanpierre E, Rauch A, Labreuche J, Susen S; Lille ICU Haemostasis COVID-19 Group. Pulmonary Embolism in Patients With COVID-19: Awareness of an Increased Prevalence. Circulation. 2020 Jul 14;142(2):184-186. doi: 10.1161/CIRCULATIONAHA.120.047430. Epub 2020 Apr 24. No abstract available. PMID 32330083